CLINICAL TRIAL: NCT02158130
Title: Effects of Aerobic Exercise Detraining on Energy Balance in Overweight Persons
Brief Title: Effects of Aerobic Exercise Detraining
Acronym: E-Mechanic_Fol
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, John Apolzan, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2014-028
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Motor Activity; Body Weight; Obesity
Keywords: Physical Inactivity; Aerobic Exercise Detraining; Body Weight; Energy Expenditure; Metabolic Syndrome
MeSH Terms: conditions — Motor Activity; Body Weight; Obesity; Sedentary Behavior; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Living: non exercise healthy living control group
- General Health: Exercise Group (8 KKW) One exercise group will obtain 8KKW (kcal/kg/week) over 3-4 sessions per week, which will result in each session lasting approximately 30 minutes. We will recruit 1 year post study intervention.
- Weight Loss: Exercise Group (20 KKW) Exercise group will obtain 20 KKW, perform in 4-5 sessions per week for approximately 50-70 minutes per session. We will recruit 1 year post study intervention.

SUMMARY:
The proposed study seeks to better understand the role of body weight, energy expenditure, and energy intake as mechanisms of body weight gain during detraining following aerobic exercise. It is hypothesized that participants in the higher dose exercise group will have greater body weight gain compared to the lower exercise dose and control group from wk 24 to wk 76 follow-up.

DETAILED DESCRIPTION:
Eligibility criteria include having successfully completed the main E-Mechanic study, be willing to archive blood samples and not being currently enrolled in another study that may effect body, energy intake or energy expenditure. The investigators will measure body weight, waist/hip circumference, blood pressure, body composition, physical activity, questionnaire about appetite/food intake and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* Completed the E-Mechanic study
* Be willing to archive blood samples
* Not participating in a study that would alter body weight, energy intake, or energy expenditure.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants that successfully enrolled and completed the E-Mechanic study and are not past 88 weeks study randomization.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Body Weight | Week 64 - 88 post study randomization
  Fasting body weight

SECONDARY OUTCOMES:
Energy Expenditure | Week 64 - 90 since study randomization
  Energy expenditure is calculated with the Sensewear Armband.
Energy Intake | Week 64 - 90 post study randomization
  Energy expenditure is calculated with the Sensewear Armband and furthermore, energy intake is calculated by adjusting TDEE for change in body weight following the methods used in doubly labeled water adjustment.

OTHER OUTCOMES:
Circumferences | Week 64-88 post study randomization
  Waist and hip circumferences
Blood Pressure | Week 64-88 post study randomization
Body Composition | Week 64 - 88 post study randomization
  Whole Body Scan GE iDXA (Dual energy x-ray absorptiometry)
Triglycerides | Week 64 - 88 post study randomization
Cholesterol | Week 64 - 88 post study randomization
  Total, HDL, and LDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — PBRC
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States